CLINICAL TRIAL: NCT01885312
Title: Tailored Mobile Text Messaging to Reduce Problem Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA021502-2; 1R34AA021502-01 (NIH)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol-Related Disorders; Alcohol Use Disorders; Alcohol Drinking; Alcoholism; Alcohol Abuse
Keywords: Drinking; Heavy Drinking; Technology; Mobile Phone; Text Message; Problem Drinking; Alcohol Problems; Alcoholism; Moderation-Oriented Treatment; Controlled Drinking; Reduced Drinking
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tailored not adaptive based Intervention (Active Comparator): Tailored Text Messaging - not adaptive in the moment and once a day intervention to reduce problem drinking
  Interventions: Behavioral: Tailored, not adaptive, based Intervention
- Ecological Momentary Assessment (Other): Mobile Assessment only
  Interventions: Other: Assessment only
- Tailored Adaptive Text Messaging (Experimental): Tailored Adaptive Text Messaging intervention to reduce problem drinking
  Interventions: Behavioral: Adaptive Tailored Intervention
- Consequence based text messaging (Active Comparator): Consequence based Text Messaging intervention to reduce problem drinking
  Interventions: Behavioral: Consequence-based Intervention

INTERVENTIONS:
Behavioral: Adaptive Tailored Intervention — Adaptive
  Arms: Tailored Adaptive Text Messaging
Behavioral: Consequence-based Intervention — Loss Framed
  Arms: Consequence based text messaging
Behavioral: Tailored, not adaptive, based Intervention — Baseline tailored not adaptive
  Arms: Tailored not adaptive based Intervention
Other: Assessment only — EMA only
  Arms: Ecological Momentary Assessment

SUMMARY:
This study is designed to develop and test a tailored adaptive text messaging/short message service (SMS) intervention for individuals interested in stopping or reducing their alcohol consumption; and test and compare it to tailored but static, once a day messaging, gain framed messaging, and ecological momentary assessment only.

DETAILED DESCRIPTION:
The proposed development study entitled, Tailored Mobile Text Messaging to Reduce Problem Drinking is designed to develop and test a tailored adaptive text messaging/short message service (SMS) intervention for individuals interested in stopping or reducing their alcohol consumption. This intervention includes messages tailored to baseline assessment results (including drinking times) that are adaptive to ongoing drinking patterns and goal achievement via interactive ecological momentary assessment (EMA). Other features include participant initiated help messaging and support network alerts. We will conduct beta research with 40 problem drinkers to assess messaging preferences and acceptability, and then conduct a pilot test with 10 PDs. In Stage 1b, we aim to test this intervention and understand the mechanisms of action of different text messaging interventions with 200 problem drinkers over a 12-week period. We propose to compare four types of messaging: 1) Tailored content and timed messaging adaptive to the participants current state (Stage 1a intervention); 2) Tailored content messaging (not adaptive or timed) sent at 3 pm every day; 3) Untailored consequence based messages sent at 3 pm every day; and 4) Brief feedback and EMA only. Assessments will be completed at baseline, through weekly EMA via SMS and at week 12 via a web-based follow-up assessment. Primary outcomes include drinks per drinking day, days of heavy drinking, and average drinks per week as measured through weekly EMA. Additional outcomes will include drinking related consequences, goal commitment and intervention satisfaction. Outcomes will be used to modify the intervention and to prepare for a larger Stage 1c RCT.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* be fluent and able to read in English at the eighth grade level
* be between the ages of 21 and 65
* have an estimated average weekly consumption of greater than 15 or 24 standard drinks per week for women and men, respectively
* be willing to reduce their drinking to non-hazardous levels
* be willing to provide informed consent
* own a mobile phone and have an active email address and are willing to receive and respond to up to 115 text messages total per month (average = 50)

Exclusion Criteria:

* Participants will be excluded from the study if they
* present with significant substance use or a current substance use disorder (for any substance other than alcohol, nicotine, or caffeine), which is defined as greater than once weekly use in the past month
* present with a serious psychiatric illness or suicide risk as measured by previous inpatient treatment, medications for psychosis or recent suicidality; demonstrate clinically severe alcoholism, as evidenced by physical withdrawal symptoms or a history of serious withdrawal symptoms (e.g., hallucinations, seizures, or delirium tremens), and score greater than 12 on the Short Alcohol Withdrawal Scale (SAWS)
* express a desire or intent to obtain additional substance abuse treatment while in the study
* report a medical condition that precludes drinking any alcohol; or
* demonstrate cognitive impairment as evidenced a score of less than 7 out of 10 on the consent form quiz

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Days of Heavy Drinking (DHD) | 12 weeks
Average Drinks per Week (ADW) | 12 weeks

SECONDARY OUTCOMES:
Drinking Related Consequences | 12 weeks
Goal Commitment | 12 weeks

OTHER OUTCOMES:
Intervention Satisfaction | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fred Muench, PhD, Principal Investigator — Feinstein Institute for Medical Research / North Shore-LIJ Health System
Locations (1):
- Feinstein Institute for Medical Research / North Shore-LIJ Health System, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once cleaned and published will make available